CLINICAL TRIAL: NCT00103896
Title: Connect to Protect (C2P) Partnerships for Youth Prevention Interventions: Phase II
Brief Title: Connect to Protect Partnerships for Youth Prevention Interventions: Phase II
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Other Study IDs: ATN 016b
Record Dates: First submitted 2005-02-15; First posted 2005-02-16 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2016-07

CONDITIONS: HIV Infection
Keywords: High-risk youth; HIV infected youth; Community mobilization; HIV serosurveys
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- HIV Infected Youth in Treatment/Care: HIV infected youth in treatment/care will be interviewed using Audio Computer-Assisted Self-Administered Interview ACASI technology to reveal possible venues where youth at high risk for acquiring the disease may be found (N = 20-30 individuals per ATN site).
- BVI Individuals: Additional data will be gathered on potential recruitment venues by administering a brief venue interview (BVI) to individuals who appear to be between 12 and 24 years old (N = unlimited individuals during 3-5 assessment periods per venue each lasting 5 hours).
- HIV Serosurvey Individuals: HIV Serosurvey Individuals Anonymous structured interview using ACASI technology and an anonymous HIV antibody assay will be administered to 20-30 young women at 2-3 targeted locations and 20-30 young men at 2-3 targeted locations whose HIV status is unknown (N = 160-360 individuals per ATN site)..

SUMMARY:
This is Phase II of a three stage project whose overall goals are to develop viable community-based HIV prevention interventions and to form and maintain the necessary community collaborations to support such Adolescent Trials Network (ATN) research activities.

This phase will describe specific locations within high-risk areas where youth, ages 12-24, spend time. HIV risk behaviors, social networking patterns and HIV prevalence among youth at these venues will be assessed by administering anonymous computerized interviews to eligible and willing youth. This information will be shared with community partners during scheduled working group meetings.

DETAILED DESCRIPTION:
This is Phase II of a three stage project whose overall goals are to develop viable community-based HIV prevention interventions and to form and maintain the necessary community collaborations to support such ATN research activities.

During this phase, each ATN site will gather additional information within high-risk areas and solicit community partner input to ultimately pinpoint the specific locations where at-risk youths, ages 12-24, may be recruited for interventions. This will be done by the following methods:

Venues will be identified by HIV+ youth at the ATN site by participation in an anonymous computerized interview. Site staff will then perform brief venue interviews (BVIs) at selected venues to assess the potential yield of youths 12-24 years old. Community partners will also provide the site staff with information on known high-risk venues. High-risk venues will further be identified by the results of anonymous computerized interviews and HIV assays obtained from eligible and willing youth participants at the venues. The interviews will gather information on HIV risk behaviors, social networking patterns and HIV prevalence among youths at these venues. This information will be shared with community partners during scheduled working group meetings.

ELIGIBILITY:
Inclusion Criteria:

Index Subjects:

* Documented HIV-infection
* Acquisition of HIV after age 9 years
* Verbal confirmation of 12-24 years of age
* Verbal report of having engaged in sexual activity (vaginal, anal and/or oral sex) within the past 12 months
* Ability to understand and willingness to provide informed consent/assent

BVI subjects:

* Youths who appear to be 12-24 years old

HIV Serosurvey subjects at the venues:

* Verbal confirmation of 12-24 years of age
* Verbal report of having engaged in sexual activity (vaginal, anal and/or oral sex) within the past 12 months
* Ability to understand and willingness to provide informed consent/assent

Exclusion Criteria:

* Visibly distraught and/or emotionally unstable (i.e. depressive mood, exhibiting manic, suicidal or violent behavior, etc.)
* Visibly intoxicated or under the influence of psychoactive agents
* Clinically presents as acutely ill

Ages: 12 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: HIV infected youth, ages 12 through 24 years old, in treatment/care at each of the 15 ATN sites will be interviewed using ACASI technology to reveal possible venues where youth at high risk for acquiring the HIV may be found. Individuals approached at 3-5 of these identified venues who appear to be 12 through 24 years will be offered a brief venue interview. Anonymous HIV serosurvey (ACASI and HIV-Ab assay) will be administered to 20-30 young women at 2-3 identified high-risk venues, and 20-30 young men at 2-3 identified high-risk venues, who provide verbal confirmation of being 12 through 24 years old, and whose HIV status is unknown to the site staff.
Sampling Method: Non-Probability Sample
Enrollment: 16706 (Actual)
Dates: Start 2003-09; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Ascertain specific community venues where at-risk youth can be recruited for interventions within the high-risk areas identified in the first Phase of the study | One time assessment at 10 months
  The outcome measure will be assessed using results from: (a) Phase I mapping; (b) Phase II interviews with HIV-infected youth; and (c) Phase II Brief Venue Interviews (BVIs). Input from community partners and ethnographic procedures will add critical information.
Describe HIV risk behaviors of adolescents and young adults recruited from targeted venues | One time assessment at 10 months
  The outcome measure will be assessed by conducting HIV serosurveys at each venue identified with youth whose HIV status is unknown.
Describe social networks of adolescents and young adults recruited from targeted venues | One time assessment at 10 months
  The outcome measure will be assessed by conducting HIV serosurveys at each venue identified with youth whose HIV status is unknown.
Describe HIV seroprevalence of adolescents and young adults recruited from targeted venues | One time assessment at 10 months
  The outcome measure will be assessed by conducting HIV serosurveys at each venue identified with youth whose HIV status is unknown.
Assess the characteristics of the community-researcher partnerships | One time assessment at 10 months
  The outcome measure will be assessed by conducting interviews with C2P staff and their community partners. Questionnaires will be completed by both parties and detailed documentation kept.
Assess quality of the community-researcher partnerships | One time assessment at 10 months
  The outcome measure will be assessed by conducting interviews with C2P staff and their community partners. Questionnaires will be completed by both parties and detailed documentation kept.
Assess outcomes of the community-researcher partnerships | One time assessment at 10 months
  The outcome measure will be assessed by conducting interviews with C2P staff and their community partners. Questionnaires will be completed by both parties and detailed documentation kept.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Ellen, MD, Study Chair — Johns Hopkins Medical Center; Ligia Peralta, MD, Principal Investigator — Division of Adolescent & Young Adult Medicine University of MD, Medical School; Donna Futterman, MD, Principal Investigator — Montefiore Medical Center; Marvin Belzer, MD, Principal Investigator — Childrens Hosp of Los Angeles, Division of Adolescent Medicine; Bret Rudy, MD, Principal Investigator — Children's Hospital of Philadelphia; Larry D'Angelo, MD, Principal Investigator — Children's National Research Institute; Cathryn Samples, MD, Principal Investigator — Boston Children's Hospital; Lisa Henry-Reid, MD, Principal Investigator — John H. Stroger Jr. Hospital and the CORE Center; Ana Puga, MD, Principal Investigator — Children's Diag. and Treatment Ctr of Ft. Lauderdale, FL; Lawrence Friedman, MD, Principal Investigator — University of Miami, School of Medicine, Div of Adolescent Medicine; Patricia Emmanuel, MD, Principal Investigator — University of South Florida, Peds Div of Infectious Disease; Sue Ellen Abdalian, MD, Principal Investigator — Tulane Medical Center; Linda Levin, MD, Principal Investigator — Mount Sinai Adolescent Health Center; Irma Febo, MD, Principal Investigator — University of Puerto Rico Medical Sciences Campus; Stephen A Spector, MD, Principal Investigator — UCSD Mother, Child, & Adolescent HIV Program; Rolando M Viani, MD, Principal Investigator — UCSD Mother, Child, & Adolescent HIV Program; Barbara Moscicki, MD, Principal Investigator — UCSF, Division of Adoles. Med; Coco Auerswald, MD, Principal Investigator — UCSF, Division of Adoles. Med
Locations (15):
- United States (14):
  - Childrens Hospital of Los Angeles, Los Angeles, California
  - UCSD Mother, Child & Adolescent HIV Program, San Diego, California
  - Univ of Califormia at San Francisco, San Francisco, California
  - Children's Hospital National Medical Center, Washington D.C., District of Columbia
  - Children's Diag. and Treatment Center, Fort Lauderdale, Florida
  - University of Miami, Miami, Florida
  - USF Peds Div. of Infectious Disease, Tampa, Florida
  - Stroger Hospital of Cook County, Chicago, Illinois
  - Tulane Medical Center, New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Childrens' Hospital of Boston, Boston, Massachusetts
  - Mount Sinai Medical Center, New York, New York
  - Montefiore Medical Center, Adolescent AIDS Program, The Bronx, New York
  - Children's Hopsital of Philadelphia, Philadelphia, Pennsylvania
- University Pediatric Hospital, San Juan, Puerto Rico

REFERENCES:
- See also: Website for the Adolescent Trials Network for HIV/AIDS Interventions — http://www.atnonline.org